CLINICAL TRIAL: NCT03142490
Title: Acupuncture as a Complementary Therapy for Infertile Patients on Treatment With in Vitro Fertilization: a Randomized Controlled Clinical Trial
Brief Title: Acupuncture as a Complementary Therapy for in Vitro Fertilization Patients: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Rubens Lene Carvalho Tavares, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60852116.2.0000.5149
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Acupuncture; Quality of Life; Infertility; Stress; Anxiety
Keywords: Acupuncture; Infertility; In vitro fertilization; Quality of life; Stress; Anxiety
MeSH Terms: conditions — Infertility; Anxiety Disorders | interventions — Acupuncture Therapy; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: In vitro fertilization patients will be randomized into two groups: treatment group (with complementary acupuncture) and control group (without complementary acupuncture).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): In vitro fertilization patients submitted to acupuncture as a complementary therapy. Patients in both groups will be evaluated by 4 different questionnaires.
  Interventions: Other: Acupuncture; Other: Questionnaires
- Control (Active Comparator): In vitro fertilization patients not submitted to acupuncture as a complementary therapy. Patients in both groups will be evaluated by 4 different questionnaires.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Acupuncture — Acupuncture as a complementary therapy will be done in In vitro fertilization patients of the treatment group.
  Arms: Treatment
Other: Questionnaires — Patients in both groups will be evaluated by 4 different questionnaires (before and after 8 to 12 weeks)

SUMMARY:
This is an open-label randomized controlled trial of the use of acupuncture in infertile patients receiving In Vitro Fertilization (IVF). Patients will be randomized into two groups: treatment group will receive acupuncture as a complementary approach to IVF and control group will receive the IVF treatment. Groups will be compared with the World Health Organization quality of life (WHOQOL-Bref), short-form 36 (SF-36), State Trait Anxiety Inventory (STAI) and Scope-Stress questionnaires.

DETAILED DESCRIPTION:
This is an open-label randomized controlled trial of the use of acupuncture in infertile patients receiving In Vitro Fertilization (IVF). Patients will be randomized into two groups: treatment group will receive acupuncture as a complementary approach to IVF and control group will receive the IVF treatment. Groups will be compared with the World Health Organization quality of life (WHOQOL-Bref), short-form 36 (SF-36), State Trait Anxiety Inventory (STAI) and Scope-Stress questionnaires. In addition, data from medical records of infertile patients submitted to in vitro fertilization for treatment of infertility will be compared in the two different treatment groups (with and without acupuncture), such as the required dose of drugs for the treatment, number of ovarian follicles, number of oocytes captured, quality of oocytes, number of embryos, quality of embryos, pregnancy and abortion rates.

ELIGIBILITY:
Inclusion Criteria:

* female patient
* age over 18 years
* diagnosis of infertility with indication of IVF
* agreement accept to participate in the study
* signature of the consent form

Exclusion Criteria:

* history of previous contact with the acupuncture technique
* severe neurological or psychiatric disorders that make it impossible to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — participant eligibility is based on self-representation
Enrollment: 100 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | after 8 acupuncture sessions (up to 12 weeks of follow-up)
  Quality of life evaluation by the WHOQOL-Bref questionnaire

SECONDARY OUTCOMES:
Quality of life 2 | after 8 acupuncture sessions (up to 12 weeks of follow-up)
  Quality of life evaluation by the SF-36 questionnaire
Stress | after 8 acupuncture sessions (up to 12 weeks of follow-up)
  Stress evaluation by the DASS 21 questionnaire
Pregnancy rate | after 8 acupuncture sessions (up to 12 weeks of follow-up)
  To compare the pregnancy rates from infertile patient records between both groups
Quality of life 3 | after 8 acupuncture sessions (up to 12 weeks of follow-up)
  Quality of life evaluation by the FERTIQOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Tavares, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No